CLINICAL TRIAL: NCT04859816
Title: Fat Absorption and Metabolism After Roux-en-Y Gastric Bypass
Acronym: FAT-BAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Morten Gadegaard Hindsø, MD, Principal Investigator, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FAT-BAR
Record Dates: First submitted 2021-04-12; First posted 2021-04-26 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Bariatric Surgery
Keywords: fat; triglyceride; triacylglycerol; Roux-en-Y gastric bypass; malabsorption
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency; Malabsorption Syndromes | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roux-en-Y gastric bypass operated participants (Experimental): Roux-en-Y gastric bypass operated participants in weight stable phase > 1 year from surgery
  Interventions: Other: Metabolic test; Other: DXA-scan; Other: MRS; Other: Feces collection
- Control participants (Experimental): Age, sex, and BMI-matched un-operated participants.
  Interventions: Other: Metabolic test; Other: DXA-scan; Other: MRS; Other: Feces collection

INTERVENTIONS:
Other: Metabolic test — Iv and oral administration of stable isotope tracers during fasting and a high-fat liquid mixed meal
Other: DXA-scan — Dual energy X-ray Absorptiometry scan of whole-body fat
Other: MRS — Magnetic resonance spectroscopy of liver fat content
Other: Feces collection — 4-day feces collection

SUMMARY:
Using intravenous and oral administration of stable isotope tracers, we will investigate the importance of altered fat absorption and altered whole body fat metabolism for the reduced postprandial systemic TAG concentrations in non-diabetic patients in weight stable phase after RYGB.

ELIGIBILITY:
Inclusion criteria, RYGB

* Age > 18 years
* RYGB > 12 months prior to inclusion
* Weight stable (± 3 kg during the last month)
* HbA1c < 48 mmol/mol before surgery, and no history of diabetes
* HbA1c < 48 mmol/mol and fasting plasma glucose < 6.1 mmol/l at inclusion

Inclusion criteria, CON

* Age > 18 years
* No former bariatric surgery
* Weight stable (± 3 kg during the last month)
* HbA1c < 48 mmol/mol, fasting plasma glucose < 6.1, and no history of diabetes

Exclusion criteria

* Thyrotoxicosis or inadequately treated hypothyreosis
* Haemoglobin < 6.5 mmol/l at inclusion
* Pregnancy (pregnancy test in fertile woman before enrolment) or breast feeding
* Medication affecting the planned examinations which cannot be paused during the study period.
* Adherence to extreme diets with excessively high or low contributions from certain macronutrients (e.g. ketogenic diet)
* Complications restricting eating behavior (e.g. postprandial hypoglycemia, vomiting or strictures)
* MR contraindications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve of plasma triacylglycerol | 6 hours
  During a high-fat liquid mixed meal test

SECONDARY OUTCOMES:
Recovery of oral stable triacylglycerol isotope tracer in feces | 4 days
  An oral stable triacylglycerol isotope tracer will be administered during a high-fat liquid mixed meal test. Feces will be collected the following 4 days to determine the recovery of the tracer in feces.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No